CLINICAL TRIAL: NCT06165107
Title: Obesity and Stroke: Exploring the Clinical Connection Through Epidemiology and Molecular Medicine
Brief Title: The Association Between Obesity-Related Indicators and Adverse Outcomes in Ischemic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Qin Zhang (Other)
Responsible Party: Sponsor-Investigator, Qin Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20230830
Record Dates: First submitted 2023-12-03; First posted 2023-12-11 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Stroke, Ischemic
Keywords: stroke; Fat; Obesity; Metabolic syndrome
MeSH Terms: conditions — Ischemic Stroke; Stroke; Platelet Glycoprotein IV Deficiency; Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ischemic stroke: We retrospectively gathered information on patients admitted for acute first-ever ischaemic stroke between January 2018 and January 2022. The following individuals were excluded from the study: 1) Those under 18 years of age; and 2) Pregnant women.
  The variables gathered included the primary test parameters of patients within 24 hours of admission, encompassing age, gender, smoking and alcohol consumption status, arterial blood pressure, fat-related indicators, comorbidities, and the primary treatments administered within the initial 24 hours.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study encompasses two cohorts: a retrospective cohort derived from a genuine clinical environment and a national multicenter prospective cohort for secondary analysis. Initially, a retrospective cohort study was conducted to investigate the impact of metabolic syndrome on the prognosis of stroke patients. Following this, a prospective cohort study was conducted to examine the relationships among metabolic syndrome, potential causative molecules, and adverse outcomes in stroke patients, as previously reported(Annals of Neurology 2011, 70(2):265-273; Lipids in Health and Disease 2024, 23(1)). Additionally, the study explored potential mediating effects among these factors. The study population comprised patients experiencing acute first-ever ischemic stroke, with diagnostic criteria established according to the International Classification of Diseases, Ninth Revision. All subjects presented conclusive neuroimaging evidence, including head computed tomography and/or magnetic resonance imaging, which was reviewed by two or more experienced neuroradiologists. Adverse outcomes were characterized as compliant endpoint events, including mortality and recurrences. The primary outcome was adverse outcomes, while the secondary outcome was recurrence-free survival (RFS).

DETAILED DESCRIPTION:
Clinical data for the derivation cohort were acquired from three medical facilities: Tongji Hospital Sino-French New City Branch in Caidian District, Tongji Hospital Qiaokou Branch in Hankou District, and Tongji Hospital Optics Valley Branch in Wuhan East Lake High-Tech Development Zone. The clinical data were sourced from the electronic medical records of Tongji Hospital, the largest healthcare facility in the Hubei region of China. Its comprehensive electronic medical record system comprises over 60 million medical records spanning from 1980 to the present. We retrospectively gathered information on patients admitted for acute first-ever ischaemic stroke between January 2018 and January 2022. The following individuals were excluded from the study: 1) Those under 18 years of age; and 2) Pregnant women.

The variables gathered included the primary test parameters of patients within 24 hours of admission, encompassing age, gender, smoking and alcohol consumption status, arterial blood pressure, fat-related indicators, comorbidities, and the primary treatments administered within the initial 24 hours.

A national multicentre prospective cohort was utilized as the validation cohort for the previous prospective study, wherein comprehensive details regarding inclusion/exclusion criteria and study implementation have been previously documented (Annals of Neurology 2011, 70(2):265-273; Lipids in Health and Disease 2024, 23(1)). The primary institutions involved in this project include: five tertiary cardiovascular institutions in China: Fuwai Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College (Beijing); The First Affiliated Hospital of Xi'an Jiaotong University (Xi'an); Tongji Hospital, Huazhong University of Science and Technology (Wuhan); Tianjin Cardiovascular Institute (Tianjin); and Daping Hospital, Army Medical University (Chongqing). Data were collected from participants in a prospective cohort study carried out from November 2000 to November 2001 at five research centers in Wuhan, Xi'an, Beijing, Tianjin, and Chongqing in China.

This prospective cohort comprised 1268 patients experiencing their first-ever stroke, with a median follow-up duration of 5 years (range, 4-5.5 years). Individuals with concurrent chronic kidney disease or chronic respiratory ailments were excluded from the study. Blood samples were collected from these patient's post-acute stroke phase (within 1 month to 1 year after onset). Upon collection, the samples were promptly placed in pre-cooled centrifuge tubes and centrifuged under controlled temperatures to separate clear plasma from cellular precipitates. Subsequently, the samples were stored in an ultra-low temperature freezer at -80 degrees Celsius. The plasma KLK1 levels were quantified using a double antibody sandwich biotin affinity enzyme-linked immunosorbent assay kit. Secondary analyses were conducted using the clinical data, with detailed descriptions of the sample collection and assay protocols outlined in previous publications(Annals of Neurology 2011, 70(2):265-273; Lipids in Health and Disease 2024, 23(1)).

ELIGIBILITY:
Inclusion Criteria:

Patients experiencing their first-ever stroke. Cases of spontaneous intracerebral hemorrhage (ICH) or ischemic stroke (IS). Patients who underwent head computed tomography and/or cranial magnetic resonance imaging within 24 hours of symptom onset.

Diagnosis of metabolic syndrome (MetS) according to the criteria established by the Chinese Diabetes Society (CDS) in 2004.

Exclusion Criteria:

Individuals under 18 years of age. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study encompasses two cohorts: a retrospective cohort derived from a genuine clinical environment and a national multicenter prospective cohort. Initially, a retrospective cohort study was conducted to investigate the impact of metabolic syndrome on the prognosis of stroke patients. Following this, a prospective cohort study was conducted to examine the relationships among metabolic syndrome, potential causative molecules, and adverse outcomes in stroke patients, as previously reported(Annals of Neurology 2011, 70(2):265-273; Lipids in Health and Disease 2024, 23(1)).
Sampling Method: Non-Probability Sample
Enrollment: 18374 (Actual)
Dates: Start 2000-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 10 years
  Death
Mortality | 5 years
  Death
Recurrence | 10 years
  Recurrent stroke
Recurrence | 5 years
  Recurrent stroke

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Ran, phd, Principal Investigator — ranxiao1001@tjh.tjmu.edu.cn
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China